CLINICAL TRIAL: NCT04791072
Title: Effectiveness of Pulmonary Rehabilitation With Tele-coaching in Patients With COVID-19
Brief Title: Tele-coaching in Patients With COVID-19
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Izmir Katip Celebi University (Other)
Responsible Party: Principal Investigator, Ilknur Naz, Assoc. Prof., Izmir Katip Celebi University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IKCSS
Record Dates: First submitted 2021-02-27; First posted 2021-03-10 (Actual); Last update posted 2021-03-10 (Actual); Status verified 2021-03

CONDITIONS: Covid19; Rehabilitation
Keywords: covid19; rehabilitation; telecoaching
MeSH Terms: conditions — COVID-19 | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Telecoaching group (Experimental): They will be given breathing exercise training and will be asked to do it every day for 8 weeks. In addition to breathing exercises, the use of incentive spirometry and aerobic exercise training will be provided. They will be asked to do breathing exercises, use of incentive spirometry and strengthening exercises for at least 20 minutes every day and 5 times a week. They will be called by phone once a week and encouraging speeches will be made.
  Interventions: Other: Exercise
- Control Group (Active Comparator): They will be given breathing exercise training and will be asked to do it every day. In addition to breathing exercises, the use of incentive spirometry and aerobic exercise training will be provided. They will be asked to do breathing exercises, use of incentive spirometry and strengthening exercises for at least 20 minutes every day and 5 times a week. There will be no interviews in the control group.
  Interventions: Other: Exercise

INTERVENTIONS:
Other: Exercise — Breathing exercise training Use of incentive spirometry Aerobic exercise training Strengthening exercises

SUMMARY:
Respiratory exercise training and aerobic exercise training will be given to patients who have been hospitalized in intensive care due to COVID 19 and underwent IMV, who were hospitalized in the service and underwent NIMV or high-flow oxygen inhalation, and whose respiratory symptoms persist after discharge. The patients in the study group will be called by phone once a week and a motivating conversation will be made. No control will be made to the control group. Before and after the training, 6-minute walking test, MRC dyspnea scale, SGRQ quality of life questionnaire and hospital anxiety depression scale will be applied.

DETAILED DESCRIPTION:
Some of the patients with COVID 19 pneumonia still have respiratory symptoms despite being treated. It has been reported that pulmonary rehabilitation programs applied in various models and in a small number to relieve or reduce these symptoms reduce dyspnea, increase exercise capacity and improve quality of life. There is no study reporting the results of a pulmonary rehabilitation program applied to COVID 19 patients in our country. The main purpose of this study is to determine the efficacy of pulmonary rehabilitation applied by telecoach to patients with severe COVID 19 pneumonia or persistent respiratory symptoms. Secondly, it is aimed to present the data of Turkish society to the literature. In accordance with this purpose investigators planed a randomised control clinical study. In our study respiratory exercise training and aerobic exercise training will be given to patients who have been hospitalized in intensive care due to COVID 19 and underwent IMV, who were hospitalized in the service and underwent NIMV or high-flow oxygen inhalation, and whose respiratory symptoms persist after discharge. The patients in the study group will be called by phone once a week and a motivating conversation will be made. No control will be made to the control group. Before and after the training, 6-minute walking test, MRC dyspnea scale, SGRQ quality of life questionnaire and hospital anxiety depression scale will be applied.

ELIGIBILITY:
Inclusion Criteria:

* Being treated in intensive care unit due to COVID-19 pneumonia,
* Receiving IMV, NIMV, or high-flow oxygen therapy
* Patients whose respiratory symptoms persist despite discharge

Exclusion Criteria:

* Patients with PCR test +
* Patients without any complaints.
* Patients who are hospitalized and discharged within 10 days
* Patients with orthopedic, neurological, cognitive problems

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2021-03-01 (Estimated); Primary Completion 2021-03-01 (Estimated); Study Completion 2021-03-01 (Estimated)

PRIMARY OUTCOMES:
Exercise Capacity | Change from baseline six minute walk distance at 8 week
  Six Minute- walk test

SECONDARY OUTCOMES:
Dyspnea Assessment | Change from baseline dyspnea at 8 week
  Medical Research Council Scale(MRC); the MRC dyspnea scale is a questionnaire that consists of five statements about perceived breathlessness. (min 1- max 5 point) Higher scores mean a worse outcome.
Quality of Life Assessment | Change from baseline quality of life at 8 week
  St. George Respiratory Questionnaire; Scores range from 0 to 100, with higher scores indicating more limitations.
Anxiety and Depression | Change from baseline anxiety and depression at 8 week
  Hospital Anxiety and Depression (HAD); The HADS questionnaire has seven items each for depression and anxiety subscales. Scoring for each item ranges from zero to three, with three denoting highest anxiety or depression level. A total subscale score of >8 points out of a possible 21 denotes considerable symptoms of anxiety or depression.

REFERENCES:
- [Derived] Sahin H, Naz I, Karadeniz G, Sunecli O, Polat G, Ediboglu O. Effects of a home-based pulmonary rehabilitation program with and without telecoaching on health-related outcomes in COVID-19 survivors: a randomized controlled clinical study. J Bras Pneumol. 2023 Jan 23;49(1):e20220107. doi: 10.36416/1806-3756/e20220107. eCollection 2023. PMID 36700571